CLINICAL TRIAL: NCT01947504
Title: Acute and Brief Intervention Following Mild Traumatic Brain Injury: A Randomized Controlled Clinical Trial
Brief Title: Early Intervention Following Mild TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elaine De Guise (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor-Investigator, Elaine De Guise, Assistant professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3525; MUHC (Other: MUHC)
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- education and support intervention (Experimental): education and support intervention
  Interventions: Behavioral: education and support intervention
- waiting list (No Intervention): waiting list and regular medical follow-up

INTERVENTIONS:
Behavioral: education and support intervention
  Arms: education and support intervention

SUMMARY:
The objective of the study is to implement and measure the efficiency of a standardized acute and brief non-pharmacological intervention (Cognitive interventions on Sleep - Anxiety - Attention - Memory) following mild TBI and observe their impact pre- and post-treatments. The ultimate goal is to have patients be re-integrated to their activities faster with lesser symptoms and have patients present lesser post-concussive symptoms. Specific objectives: 1) Measure the effect of an acute and brief non-pharmacological intervention on PCS symptoms, sleep, headaches, affect, cognition and functional outcome following mild TBI; 2)To redefine a model of outcome prediction following mild TBI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild TBI

Exclusion Criteria:

* Psychiatric diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Recurrence of post-concussive symptoms | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Audrit H, Beauchamp MH, Tinawi S, Lague-Beauvais M, Saluja R, de Guise E. Multidimensional Psychoeducative and Counseling Intervention (SAAM) for Symptomatic Patients With Mild Traumatic Brain Injury: A Pilot Randomized Controlled Trial. J Head Trauma Rehabil. 2021 Jul-Aug 01;36(4):E249-E261. doi: 10.1097/HTR.0000000000000653. PMID 33656475